CLINICAL TRIAL: NCT05053191
Title: Advancing Family-Centered Care Nursing Practices in Inpatient Oncology Care
Brief Title: Advancing Nursing Practices in Hospital Oncology Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-448
Record Dates: First submitted 2021-09-14; First posted 2021-09-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Cancer; Gastrointestinal Disease; Nurse's Role
Keywords: Family Caregiver; Family Centered Care; Inpatient Oncology Care; Nursing Practices; 20-448; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurses (Experimental): MSKCC day-shift nurses (Clinical Nurse I to IV) assigned to the GI inpatient unit (MH16) at the time of study, all of whom provide initial and ongoing assessment of patients' physical, psychosocial, cultural and informational needs
  Interventions: Behavioral: Partnership, Assessment, Care and Transition training intervention

INTERVENTIONS:
Behavioral: Partnership, Assessment, Care and Transition training intervention — Partnership, Assessment, Care and Transition to psychosocial resources. Nurses who participate in PACT will receive 8 hours of training in a single, full-day workshop. We will train nurses in clusters of 10-12 nurses at one time, which will allow for cross-coverage with minimal disruption to workflow, and provide a more intimate, small-group learning environment.
  Other Names: PACT

SUMMARY:
The purpose of this study is to find out if a new training program for nurses called PACT (Partnership, Assessment, Care, and Transition) will be effective and relevant in helping nurses gain the skills needed to provide high-quality family-centered care. Family-centered care skills include engaging family caregivers as partners in patient care, and strengthening their capacity for caregiving by assessing family support needs and facilitating access to resources when needed. The study will also look at whether the quality of nurses' family-centered care skills is associated with improved outcomes for family caregivers. Both nurses and family caregivers will be enrolled in this study. Participants will be nurses/caregivers who care for advanced GI cancer patients admitted to Memorial Sloan Kettering.

ELIGIBILITY:
Inclusion Criteria:

Nurses:

* MSKCC day-shift nurses and/or night-shift nurses (Clinical Nurse I to IV) assigned to the GI inpatient unit (M16) at the time of study, all of whom provide initial and ongoing assessment of patients' physical, psychosocial, cultural and informational needs
* Nurse is comfortable speaking and reading English as per self report

Family caregivers (FC) - Phase 1b:

* Adult (≥18 yrs) family caregiver (family caregiver is defined here as any informal caregiver who is a relative, friend or legal representative) who self-identifies and/or is identified by the nursing staff as involved in the care of an MSK cancer patient who either:

  * is currently admitted to the M16 unity for at least 12 hours OR
  * has been discharged from the M16 unit within the last 2 weeks
* English-speaking as per self-report
* Only one FC per patient case will be invited to participate.

M16 Patients (chart review only):

* Adult (≥18 yrs) cancer patient who is currently admitted in the M16 unit at Memorial Hospital for at least 12 hours o English speaking as per self-report

Exclusion Criteria:

Nurses:

* Nurse plans to leave MSK or the GI unit within 3 months as per self-report
* [Phases 2-4] Nurse refuses observation of consultations as per self-report

Family caregivers (FC) - Phase 1b:

* FC's patient is deceased at time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of nurses' use of family centered care practices | 30 days
  Frequency of nurses' use of family centered care practices as observed during inpatient consultations with family caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Talia Zaider, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org